CLINICAL TRIAL: NCT06433596
Title: Effectiveness and Safety of Autologous Plasma Rich in Platelets and Focal Shock Waves for the Erectile Dysfunction Treatment
Brief Title: Autologous PRP and Focal Shock Waves for Erectile Dysfunction
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Elexial Research Limited (Other)
Collaborators: Boston Medical Group (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PRP-SW-03; 2022-002985-34 (EudraCT Number)
Record Dates: First submitted 2024-05-23; First posted 2024-05-29 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2025-08

CONDITIONS: Erectile Dysfunction
Keywords: Erectile dysfunction; Platelet-rich plasma; Shock wave therapy; Randomized clinical trial
MeSH Terms: conditions — Erectile Dysfunction

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Autologous PRP (Experimental): 3 injections of 10 cc of autologous Platelet Rich Plasma (PRP) + 6 sessions of placebo shock waves
  Interventions: Other: Platelet-rich plasma; Other: Sham shock waves therapy
- Combined therapy (Experimental): 3 injections of 10 cc of autologous PRP + 6 sessions of focal shock waves.
  Interventions: Other: Platelet-rich plasma; Other: Shock waves therapy
- Placebo control (Placebo Comparator): 3 injections of 10 cc of saline solution + 6 sessions of placebo shock waves
  Interventions: Other: Placebo PRP; Other: Sham shock waves therapy
- Shock waves (Active Comparator): 3 injections of 10 cc of saline solution + 6 sessions of waves of focal shock.
  Interventions: Other: Shock waves therapy; Other: Placebo PRP

INTERVENTIONS:
Other: Platelet-rich plasma — 3 injections of 10 cc of autologous Platelet Rich Plasma (PRP), weeks 1, 5 and 9
  Other Names: PRP
  Arms: Autologous PRP; Combined therapy
Other: Shock waves therapy — 6 sessions of focal shock waves, 1 per week
  Arms: Combined therapy; Shock waves
Other: Placebo PRP — 3 injections of 10 cc of saline solution, weeks 1, 5 and 9
  Arms: Placebo control; Shock waves
Other: Sham shock waves therapy — 6 sessions of sham shock waves, 1 per week
  Other Names: Placebo therapy
  Arms: Autologous PRP; Placebo control

SUMMARY:
The goal of this clinical trial is to learn if Platelet-rich plasma (PRP) combined with Shock-wave therapy (SWT) works to treat moderate or mild to moderate erectile dysfunction. It will also learn about the safety of this combined therapy.

The main questions it aims to answer are:

* Does Combined therapy PRP + SWT improve erection in men with moderate or mild to moderate erectile dysfunction?
* What medical problems do participants have when receiving Combined therapy PRP + SWT?

Researchers will compare Combined therapy PRP + SWT to placebo therapy (a look-alike substance that contains no PRP) to see if Combined therapy PRP + SWT works to treat moderate or mild to moderate erectile dysfunction.

Participants will:

* Take a lab test to evaluate their platelets
* Answer some questionnaires to assess your erectile function
* Receive Combined therapy PRP + SWT (3 sessions PRP + 6 sessions SWT) or placebo therapy for 9 weeks
* Visit the clinic one month, 3 months, and 6 months after finishing the treatment for checkups and tests

DETAILED DESCRIPTION:
The goal of this clinical trial is to evaluate the effectiveness of intracavernosal autologous platelet-rich plasma therapy, compared with placebo, for the treatment of moderate or mild to moderate erectile dysfunction, measured as improvement in the IIEF-EF questionnaire score.

Study design: Randomized, double-blind, placebo-controlled clinical trial, phase III. The study will include four groups:

* G1 - Autologous PRP: Autologous Platelet Rich Plasma (PRP) + placebo shock waves
* G2 - combined therapy: Autologous PRP + focal shock waves
* G3 - placebo control: Placebo PRP + placebo shock waves
* G4 - shock waves: PRP placebo + shock waves

  116 subjects will be included, who will be randomized in a 1:1:1:1 ratio in the four groups described above.

The change in the International Index of Erectile Function - Erectile Function domain (IIEF-EF) score, the change in the Erection Hardness Score (EHS), and the adverse events will be evaluated at the end of treatment, and 1, 3, and 6 months of follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Men over 18 years of age.
2. Erectile dysfunction present for more than 3 months in more than 50% of intercourse.
3. Baseline score of the IIEF-EF questionnaire between 11 and 21.
4. Stable heterosexual relationship of at least 6 months.
5. Commitment to have at least 3 vaginal sexual relations per month after completing treatment.
6. Commitment not to use other natural, oral, or intracavernous pharmacological treatments during the treatment and up to 6 months after its completion.
7. A patient who agrees to voluntarily enter the study by signing an informed consent.

Exclusion Criteria:

1. Score of 4 on the EHS scale.
2. Patients with an international normalized ratio (INR) greater than 3.
3. Patients with sickle cell anemia.
4. Patients with clinical suspicion of hypogonadism (ADAM positive).
5. Acromegaly, gigantism, Addison disease, hyperprolactinemia, androgen deficiency.
6. Active bladder, prostate, or colon cancer.
7. Radical prostatectomy or other radical pelvic surgery.
8. History of pelvic radiotherapy.
9. Spinal cord injury or other neurological disease associated with erectile dysfunction.
10. Penile anatomical dysfunction, penile implant.
11. Platelet diseases or coagulation disorders.
12. Treatment with oral anticoagulants.
13. Platelet count outside the normal range (150 to 400 × 109/L).
14. Patients with active infections or lesions of the penis or pubic area.
15. Patients with erectile dysfunction secondary to drug treatment (antiandrogen therapy, Alpha-blockers for benign prostatic hyperplasia, use of corticosteroids, antiparkinsonian drugs, antipsychotics).
16. Patients with erectile dysfunction of psychological origin.
17. Abuse of psychoactive substances (including alcohol).
18. Cognitive or physical illness that prevents you from participating in the study, self-filling out the questionnaires, or attending therapies and controls.
19. Inability to attend therapies and controls.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — The participant must be male by biological sex and their gender identity must be male
Enrollment: 116 (Estimated)
Dates: Start 2024-05-06 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in IIEF-EF score | From enrollment to the third month of follow-up at 21 weeks
  Change in International Index of Erectile Function - Erectile Function domain (IIEF-EF) score between baseline and week 21 (3 months after completion of treatment)

SECONDARY OUTCOMES:
Change in IIEF-EF score 1- month follow-up | From enrollment to the first month of follow-up at 13 weeks
  Change in International Index of Erectile Function - Erectile Function domain (IIEF-EF) score between baseline measurement and measurement at week 13
Change in IIEF-EF score 6 months follow-up | From enrollment to the sixth month of follow-up at 33 weeks
  Change in IIEF-EF score between baseline measurement and measurement at week 33
Minimum clinically significant difference | From enrollment to the first, third and sixth month of follow-up at 13, 21, and 33 weeks
  Proportion of patients achieving the minimum clinically significant difference in the IIEF-EF score (5 points)
Change in Erection Hardness Score (EHS) | From enrollment to the first, third and sixth month of follow-up at 13, 21, and 33 weeks
  Change in EHS between baseline measurement and measurement at weeks 13, 21, and 33
Ability to penetrate | From enrollment to the first, third and sixth month of follow-up at 13, 21, and 33 weeks
  Proportion of patients who accomplish to penetrate after treatment, evaluated by the change in the EHS from 1 or 2 at baseline to 3 or 4 in weeks 13, 21 and 33.
Quality of sexual life | From enrollment to the first, third and sixth month of follow-up at 13, 21, and 33 weeks
  Change in the score of the sexual quality of life questionnaire (SLQQ) between the baseline measurement and the measurement at weeks 13, 21 and 33.
Global assessment | From enrollment to the first, third and sixth month of follow-up at 13, 21, and 33 weeks
  Change in the score of the global assessment questionnaire (GAQ) at weeks 13, 21 and 33.
Adverse events incidence | From the first intervention to end of follow-up at 33 weeks
  Incidence of PRP-related adverse events during the study

CONTACTS AND LOCATIONS:
Overall Officials: Jose Benitez, MD, Principal Investigator — Boston Medical Group
Locations (1):
- Boston Medical Group Spain S.L.U, Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data (IPD) collected throughout the trial, except personal identification data of the participants
Supporting Information: Study Protocol, CSR, Analytic Code
Time Frame: Beginning 1 month after publication with no end date
URL: https://www.elexialresearch.com/